CLINICAL TRIAL: NCT06362291
Title: Comparison of MRI Artificial Intelligence-guided Cognitive Fusion-targeted Biopsy Versus Routine Cognitive Fusion-targeted Prostate Biopsy in Prostate Cancer Diagnosis: a Prospective Randomized Controlled Trial
Brief Title: Comparison of MRI AI-cTB Versus Routine cTB in Prostate Cancer Diagnosis: a Prospective Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, LIU Yi, Associate chief physician, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2023IR27
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Artificial intelligence; Cognitive targeted biopsy; Diagnosis; Randomized controlled trial
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRI-AI-guided cTB (AI-cTB) group (Experimental): The trained AI algorithms were embedded into proprietary structured reporting software. Before prostate biopsy, the MR images of patients in the AI-cTB group were uploaded to the AI software. The prostate gland and suspicious lesions were annotated and highlighted by AI software. The urologists who were blinded to the picture archiving and communication system (PACS) and MRI reports read the AI findings at their discretion and then conducted 3-5 core TB at each suspicious lesion, followed by 12 core SB. If there was no suspicious lesion detected by the AI, only SB would be performed.
  Interventions: Procedure: MRI-AI guided cognitive prostate targeted biopsy
- Routine cTB group (Experimental): For patients in the cTB group, the MR images and reports were viewed by urologists preceding the biopsy. Then 3-5 core cTB were performed, followed by 12 core SB. In patients with negative MRI findings, only SB was performed. When urologists performed biopsies, ultrasound technicians and radiologists were present to provide necessary assistance.
  Interventions: Procedure: Routine cognitive prostate targeted biopsy

INTERVENTIONS:
Procedure: MRI-AI guided cognitive prostate targeted biopsy — Before prostate biopsy, the MR images of patients in the AI-cTB group were uploaded to the AI software. Then the images with suspicious lesions highlighted by AI software were viewed by urologists. Biopsies were performed under the guidance of TRUS through the transrectal or transperineal route.
  Arms: MRI-AI-guided cTB (AI-cTB) group
Procedure: Routine cognitive prostate targeted biopsy — Before prostate biopsy, the MR images and reports were viewed by urologists preceding the biopsy. Biopsies were performed under the guidance of TRUS through the transrectal or transperineal route.
  Arms: Routine cTB group

SUMMARY:
The goal of this clinical trial is to compare the cancer detection rates of MRI artificial intelligence-guided cTB (AI-cTB) and routine cTB, and explore the added value of using AI for the guidance of cTB. The main questions it aims to answer are:

Does AI-cTB promote the accurate diagnosis and treatment of prostate cancer? What's the value of prostate MRI artificial intelligence assistant diagnosis system in developing the best scheme of prostate biopsy? What's the value of prostate MRI artificial intelligence assistant diagnosis system in predicting the pathological results of prostate targeted biopsy?

Researchers will compare the cancer detection rates of AI-cTB and routine cTB to explore the added value of using AI for the guidance of cTB.

Participants will:

Receive AI-cTB or routine cTB.

DETAILED DESCRIPTION:
Cognitive fusion MRI-guided targeted biopsy (cTB) has been widely used in the diagnosis of prostate cancer (PCa). However, cTB relies heavily on the operator's experience and confidence in MRI readings. The goal of this clinical trial is to compare the cancer detection rates of MRI artificial intelligence-guided cTB (AI-cTB) and routine cTB, and explore the added value of using AI for the guidance of cTB.

The main questions it aims to answer are:

Does AI-cTB promote the accurate diagnosis and treatment of prostate cancer? What's the value of prostate MRI artificial intelligence assistant diagnosis system in developing the best scheme of prostate biopsy? What's the value of prostate MRI artificial intelligence assistant diagnosis system in predicting the pathological results of prostate targeted biopsy?

This prospective, single-institution RCT compared the csPCa detection rates of the AI-cTB and routine cTB. Participants were prospectively enrolled at Peking University First Hospital (Beijing, China) from August 2023 to July 2024. Participants were randomly allocated to AI-cTB group and routine cTB group.

Researchers will compare the cancer detection rates of AI-cTB and routine cTB to explore the added value of using AI for the guidance of cTB.

Participants will:

Receive AI-cTB or routine cTB.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the patient is between 45 and 85.
2. Patients with complete multiparametric magnetic resonance imaging (mpMRI) data of Peking University First Hospital, qualified image quality control, suspicious lesions, and Prostate Imaging Reporting and Data System version 2.1 (PI-RADS V2.1) of ≥ 3.
3. Patients were in accordance with the indication of prostate biopsy, including patients with suspicious prostate nodes found by digital rectal examination (DRE), the suspicious lesions found by transrectal ultrasound (TRUS) or MRI, total prostate-specific antigen (tPSA) >10ng/mL, tPSA 4-10ng/mL with free-to-total PSA ratio (f/tPSA) <0.16 or PSA density (PSAD) >0.15.
4. Patients were in accordance with the indication of repeated prostate biopsy (patients with atypical acinar hyperplasia or high-grade intraepithelial neoplasia, especially when the pathological results of multi-needle puncture were as above; re-examination of PSA > 10 ng/ml; re-examination of PSA 4~10ng/ml, abnormal f/tPSA, abnormal PSAD, abnormal DRE, or imaging abnormalities; for patients with the results of re-examination of PSA 4~10ng/ml and with close follow-up, PSA for 2 consecutive years > 10ng/ml or PSA volume > 0.75/ml/ years). The time interval between the two prostate biopsies should be longer than three months.
5. The targeted prostate biopsy pathological results of above lesions were complete. The time interval between targeted prostate biopsy and prostate mpMRI examination should not exceed one month.
6. Patients with complete clinical information.

Exclusion Criteria:

1. The mpMRI data was unqualified or incomplete.
2. Patients had received radiotherapy, chemotherapy, androgen deprivation therapy, or surgery treatment before prostate mpMRI examination or prostate biopsy.
3. The mpMRI of Peking University First Hospital did not find suspicious prostate lesions.
4. Patients were not in accordance with the indication of prostate biopsy or were not received systematic biopsy combined with targeted biopsy.
5. The patient could not cooperate to complete the systematic biopsy combined with targeted biopsy. The patients or their family members refused to participate in this study.
6. Patients with incomplete clinical information.

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
The clinically significant prostate cancer (csPCa) detection rate for targeted biopsy (TB) and TB combined with systematic biopsy (SB) | One month after the biopsy procedure.
  csPCa was defined as PCa with a grade group > 2 or GS ≥ 7. The reference standard was the pathological results of the combination of TB (AI-cTB or cTB) and SB.

SECONDARY OUTCOMES:
The PCa detection rate | One month after the biopsy procedure.
  The PCa detection rate for targeted biopsy (TB) and TB combined with systematic biopsy (SB)
The Gleason score (GS) of the biopsy sample | One month after the biopsy procedure.
  The Gleason score was reported by senior uropathologists according to the Standards of Reporting for MRI Targeted Biopsy Studies (START) criteria and interpreted according to the recommendations of the International Society of Urological Pathology (ISUP) Grade Group.
The GS of radical prostatectomy (RP) specimens | One month after the biopsy procedure.
  The overall grade was assigned based on the part with the highest Gleason score according to the recommendations of the ISUP.

CONTACTS AND LOCATIONS:
Overall Officials: Yi LIU, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Deng R, Liu Y, Wang K, Ruan M, Li D, Wu J, Qiu J, Wu P, Tian P, Yu C, Shang J, Zhao Z, Zhou J, Cai L, Wang X, Gong K. Comparison of MRI artificial intelligence-guided cognitive fusion-targeted biopsy versus routine cognitive fusion-targeted prostate biopsy in prostate cancer diagnosis: a randomized controlled trial. BMC Med. 2024 Nov 13;22(1):530. doi: 10.1186/s12916-024-03742-z. PMID 39533250